CLINICAL TRIAL: NCT06984341
Title: A Phase I, Multicenter, Open-label Study to Evaluate the Safety, Tolerability, Cellular Kinetics, Pharmacodynamics, and Efficacy of P-CD19CD20-ALLO1 in Patients With Severe, Treatment-refractory Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Safety, Tolerability, Cellular Kinetics, Pharmacodynamics, and Efficacy of P-CD19CD20-ALLO1 in Participants With Severe, Treatment-refractory Systemic Lupus Erythematosus (SLE)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GA45767
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus Nephritis; CAR-T therapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): Participants with SLE (with or without LN) will receive the following interventions and dose escalated per protocol:
  Biological: P-CD19CD20-ALLO1 Drug: Cyclophosphamide Drug: Fludarabine Drug: Rimiducid
  Interventions: Biological: P-CD19CD20-ALLO1 Cells; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rimiducid
- Dose Expansion (LN cohort) (Experimental): Participants with SLE (with LN) will receive the following interventions at or below the maximum tolerated dose (MTD), as determined in the dose escalation stage per protocol:
  Biological: P-CD19CD20-ALLO1 Drug: Cyclophosphamide Drug: Fludarabine Drug: Rimiducid
  Interventions: Biological: P-CD19CD20-ALLO1 Cells; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rimiducid
- Dose Expansion (ERL cohort) (Experimental): Participants with SLE (with ERL) will receive the following interventions at or below the maximum tolerated dose (MTD), as determined in the dose escalation stage per protocol:
  Biological: P-CD19CD20-ALLO1 Drug: Cyclophosphamide Drug: Fludarabine Drug: Rimiducid
  Interventions: Biological: P-CD19CD20-ALLO1 Cells; Drug: Cyclophosphamide; Drug: Rimiducid

INTERVENTIONS:
Biological: P-CD19CD20-ALLO1 Cells — P-CD19CD20-ALLO1 cells will be administered intravenously as per the schedule specified in the protocol.
Drug: Cyclophosphamide — Cyclophosphamide will be administered intravenously.
Drug: Fludarabine — Fludarabine will be administered intravenously.
  Arms: Dose Escalation; Dose Expansion (LN cohort)
Drug: Rimiducid — Rimiducid will be used as a rescue therapy in the event of the occurrence of severe or life-threatening adverse events. It will be administered intravenously.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of P-CD19CD20-ALLO1 in participants with highly active, severe, refractory SLE with or without lupus nephritis (LN). This study includes a dose-escalation stage followed by an expansion stage. It will also evaluate the cellular kinetics (CK), pharmacodynamics (PD), and efficacy of P-CD19CD20-ALLO1.

ELIGIBILITY:
Key Inclusion criteria:

18-75 years old

SLE diagnosis per 2019 EULAR/ACR classification criteria ≥ 24 weeks

Autoantibody positive and low complement at screening

Treatment refractory: Failed ≥ 2 treatments for at least 3 months

Highly active disease:

SLEDAI-2K ≥ 8 (excluding alopecia, headache, and fever; additional protocol-specified requirements to enhance specificity of findings)

BILAG-2004 cat A in ≥ 1 organ system and/or cat B in ≥ 2 organ systems (excluding constitutional, musculoskeletal, and/or mucocutaneous organ systems for category B)

PGA score ≥ 1.0 on a 0 to 3 VAS

For patients with lupus nephritis:

Biopsy-proven Class III or IV (± Class V) active LN per 2018 ISN/RPS criteria within 12 months of screening

Modified NIH activity index ≥ 1/24

UPCR ≥ 1g/g

Key Exclusion criteria:

Participants who are pregnant, breastfeeding, or intend to become pregnant within the timeframe in which contraception is required

Prior treatment with CAR T-cell therapy, B-cell-targeting T-cell-dependent bispecific antibody, gene therapy product, total body irradiation, allograft organ transplant, or hematopoietic stem cell transplant

Significant organ impairment (renal, hepatic, cardiac, or pulmonary) or uncontrolled medical disease which, in the investigator's opinion would preclude patient participation or that may require treatment with systemic corticosteroids or immunosuppressants during the study

Active severe or unstable neuropsychiatric disease

Protocol-specified active or chronic infections, recent major episode of infection

High-risk medical conditions (e.g. high bleeding risk, history of cancer, recent major surgery, history of HLH/MAS, substance abuse within the previous year)

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2033-11-01 (Estimated); Study Completion 2033-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Toxicities (DLTs) at Each Dose Level of P-CD19CD20-ALLO1 | Day 1 up to Day 29
Number of Participants With Adverse Events (AEs) | Up to 5 years

SECONDARY OUTCOMES:
Number of Chimeric Antigen Receptor (CAR) Transgene Copies in Blood Assessed by Droplet Digital Polymerase Chain Reaction (ddPCR) | Up to 5 years
B-cell Levels in the Blood | Up to 5 years
Percentage of Participants who Achieve Sustained Drug-free Definition of Remission in SLE (DORIS) | From Week 24 through Week 52
  Drug-free DORIS is defined as a SLEDAI-2K = 0 and a PGA <0.5 (on a 3-point PGA-visual analog scale [VAS]), without corticosteroids or other immunosuppressants.
Number of Participants With Anti-CAR T Antibodies | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.

IPD SHARING:
Plan to Share IPD: No